CLINICAL TRIAL: NCT03277976
Title: Pulmonary Vein Isolation Guided by Ablation Index
Brief Title: Pulmonary Vein Isolation Guided by Ablation Index (Ablation Index Registry Study)
Acronym: AIR
Status: Completed | Type: Observational
Sponsor: Clinica Mediterranea (Other)
Responsible Party: Sponsor
Other Study IDs: AIR Study
Record Dates: First submitted 2017-07-27; First posted 2017-09-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation;; catheter ablation;; pulmonary vein isolation; ablation index
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ThermoCool SmartTouch 1: In this cohort are included patients who will undergo atrial fibrillation ablation using the ThermoCool SmartTouch Catheter and Ablation Index range: 380 for the posterior wall and 500 for the anterior wall
  Interventions: Device: PVI using ThermoCool® SmartTouch® Catheter
- ThermoCool SmartTouch 2: In this cohort are included patients who will undergo atrial fibrillation ablation using the ThermoCool SmartTouch Catheter and Ablation Index range: 330 for the posterior wall and 450 for the anterior wall
  Interventions: Device: PVI using ThermoCool® SmartTouch® Catheter
- ThermoCool SmartTouch SF 1: In this cohort are included patients who will undergo atrial fibrillation ablation using the ThermoCool SmartTouch SF Catheter and Ablation Index range: 330 for the posterior wall and 450 for the anterior wall
  Interventions: Device: PVI using ThermoCool® SmartTouch SF® Catheter
- ThermoCool SmartTouch SF 2: In this cohort are included patients who will undergo atrial fibrillation ablation using the ThermoCool SmartTouch SF Catheter and Ablation Index range: 380 for the posterior wall and 500 for the anterior wall
  Interventions: Device: PVI using ThermoCool® SmartTouch SF® Catheter

INTERVENTIONS:
Device: PVI using ThermoCool® SmartTouch® Catheter — PVI using RFA, using ThermoCool® SmartTouch® Catheter (Biosense Webster Inc., CA, US), guided by Ablation Index
  Groups: ThermoCool SmartTouch 1; ThermoCool SmartTouch 2
Device: PVI using ThermoCool® SmartTouch SF® Catheter — PVI using RFA, using ThermoCool® SmartTouch SF® Catheter (Biosense Webster Inc., CA, US), guided by Ablation Index
  Groups: ThermoCool SmartTouch SF 1; ThermoCool SmartTouch SF 2

SUMMARY:
This is a prospective, multi-center, research study designed to evaluate the acute achievement of pulmonary vein (PV) isolation with ThermoCool SmartTouch (ST) and ThermoCool SmartTouch SF (STSF) catheter using the Ablation Index Module.

DETAILED DESCRIPTION:
This is a prospective, multi-center, research study designed to evaluate the acute achievement of pulmonary vein (PV) isolation with ThermoCool SmartTouch (ST) and ThermoCool SmartTouch SF (STSF) catheter using the Ablation Index Module.

Subjects with paroxysmal and persistent atrial fibrillation (AF) will undergo catheter ablation using commercially approved devices (mapping system and catheters).

Patients will be followed up for 12 months to measure the recurrence of AF. This study is expected to start in September 2017 and to continue for approximately 26 months. It is anticipated that this study will require approximately 12 months for subject enrollment. Patients will be followed up for at least 12 months. Data analysis is expected to require approximately 2 months. At least 320 consecutive patients will be enrolled in the study centers. Patients will be divided in 4 groups and enrollment will stop when at least 80 patients will be enrolled in each group. The investigators evaluate two ablation catheters (ST and STSF) and two different ablation index settings (380 posterior - 500 anterior and 330 posterior - 450 anterior). Given that the rate of PV isolation with a standard wide antral circumferential ablation technique (WACA) is about 70%, the investigators want to test if one of two catheters or one of ablation index settings can increase the PV isolation rate of at least 10% (from 70% to 80%, 95% CI 75-85%).

Primary endpoint The primary objective of this study is to evaluate which ablation strategy increase the rate of WACA PV isolation, validated by mean of LASSO catheter, after first encirclement, from 70% to 80%.

Secondary endpoints Incidence of early PV reconnection 30 minutes after acute PV isolation. Difference in procedural and fluoroscopy time between the two groups. Incidence of AF recurrence during the blanking period (3-months after ablation).

Safety of the ablation procedure. At least 320 patients undergoing catheter ablation for paroxysmal or persistent AF will be enrolled.

Inclusion Criteria The following criteria must be met for subjects to be eligible for inclusion into the study Subject is indicated for catheter ablation for paroxysmal AF Subject is > 18 years old Subject is < 80 years old Subject is on adequate anticoagulation therapy

Exclusion Criteria The following criteria are exclusions for study participation Patients who had already undergo an AF ablation procedure Patients with left ventricular ejection fraction < 35% Women of childbearing potential who are or might be pregnant Hematological contraindications to ionizing radiation exposure Presence of complex congenital heart disease, and cardiac surgery within 1 month from enrollment

Patients will be screened in ambulatory and scheduled for AF ablation according to current guide lines. Ablation will be usually performed under effective oral anticoagulation. Anticoagulation could be withdrawn before admission, so as antiarrhythmic drugs will be removed before scheduled procedure. Patients in AF or with a CHA2DS2-VASc score ≥ 1 will undergo transesophageal echocardiography within 48 hours prior to the ablation. For all other patients transesophageal echocardiography is optional. Cardiac MRI or Cardiac CT scan could be executed as a reference for volume estimations obtained with the mapping system.

Ablation will be carried out under mild or conscious sedation, at least 2 femoral vein access will be obtained and in some patients 1 subclavian vein. One diagnostic catheter will be positioned in the coronary sinus. One or two transseptal accesses to the left atrium will be achieved using a standard approach. Then, the LASSO catheter and the ablation catheter (ST and STSF) will be placed in the left atrium. Heparin will be administered before the transseptal punctures to maintain an activated clotting time ≥ 300 seconds for the duration of the procedure. Left atrium mapping will be performed in sinus rhythm. Patients with atrial fibrillation at the beginning of the index procedure will undergo electrical cardioversion. After left atrium reconstruction the effective PV-left atrium electrical connection will be checked with LASSO. In all groups a wide antrum circumferential ablation aimed at PV isolation will be performed using contact force threshold range between 5-40 g (14), and the Ablation Index Module, with the following preset: respiration adjustment; stability range 3 mm, stability time 3 sec, force over time 25% of time, 3 g and ablation index thresholds: 500 for anterior wall and 380 for posterior wall or 450 for anterior wall and 330 for posterior wall; contiguity lesion 5-6 mm (15-16). The default power setting will be 30 W, with ranges of 20-40 W. At the end of the ablation effective PV isolation (entry and exit block), will be checked with LASSO catheter. After PV isolation will be achieved, the reconnection of the same vein will be evaluated after a 30 minute period from the initial isolation or after adenosine infusion or isoproterenol. If the vein reconnects to the atrium, the ablation will be directed to the gaps identified by the LASSO catheter. All patients will undergo a post-procedural ECG and, optional, an echocardiogram to exclude pericardial effusion or other acute complications. After ablation, patients will undertake regular follow-up assessments (scheduled at 3 months) including a detailed history, physical examination, 12-lead standard electrocardiography, and 24-h Holter monitoring. Patients who will not report any symptoms related to the previous arrhythmia during a supplementary detailed follow up (6-12 months subsequent to catheter ablation) will be considered free of arrhythmia recurrence

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for catheter ablation for paroxysmal AF;
* Subject is > 18 years old;
* Subject is < 80 years old ;
* Subject is on adequate anticoagulation therapy

Exclusion Criteria:

* Patients who had already undergo an AF ablation procedure;
* Patients with left ventricular ejection fraction < 35%
* Women of childbearing potential who are or might be pregnant
* Hematological contraindications to ionizing radiation exposure
* Presence of complex congenital heart disease, and cardiac surgery within 1 month from enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with paroxysmal and persistent atrial fibrillation (AF) will undergo catheter ablation using commercially approved devices (mapping system and catheters).
Sampling Method: Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate which ablation strategy increase the rate of WACA PV isolation, validated by mean of LASSO catheter, after first encirclement, from 70% to 80%. | From the end of the WACA PV isolation up to 5 min after

SECONDARY OUTCOMES:
Incidence of early PV reconnection 30 minutes after acute PV isolation. | Up to 30 min after the effective pulmonary vein isolation
Difference in procedural and fluoroscopy time between the two groups | From the beginning of the index procedure to the end of index procedure
Incidence of AF recurrence during the blanking period | Up to 3 months after the ablation procedure
Incidence of treatment-emergent adverse events. | Number of participants with treatment-related adverse events as assessed by CTCAE v4.0, from the index procedure to one-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Mediterranea, Naples, Italy

REFERENCES:
- [Background] El Haddad M, Taghji P, Phlips T, Wolf M, Demolder A, Choudhury R, Knecht S, Vandekerckhove Y, Tavernier R, Nakagawa H, Duytschaever M. Determinants of Acute and Late Pulmonary Vein Reconnection in Contact Force-Guided Pulmonary Vein Isolation: Identifying the Weakest Link in the Ablation Chain. Circ Arrhythm Electrophysiol. 2017 Apr;10(4):e004867. doi: 10.1161/CIRCEP.116.004867. PMID 28381417
- [Background] Das M, Loveday JJ, Wynn GJ, Gomes S, Saeed Y, Bonnett LJ, Waktare JEP, Todd DM, Hall MCS, Snowdon RL, Modi S, Gupta D. Ablation index, a novel marker of ablation lesion quality: prediction of pulmonary vein reconnection at repeat electrophysiology study and regional differences in target values. Europace. 2017 May 1;19(5):775-783. doi: 10.1093/europace/euw105. PMID 27247002
- [Result] Das M, Wynn GJ, Morgan M, Lodge B, Waktare JE, Todd DM, Hall MC, Snowdon RL, Modi S, Gupta D. Recurrence of atrial tachyarrhythmia during the second month of the blanking period is associated with more extensive pulmonary vein reconnection at repeat electrophysiology study. Circ Arrhythm Electrophysiol. 2015 Aug;8(4):846-52. doi: 10.1161/CIRCEP.115.003095. Epub 2015 Jun 24. PMID 26108982
- [Result] Stabile G, Di Donna P, Schillaci V, Di Monaco A, Iuliano A, Caponi D, Urraro F, Solimene F, Grimaldi M, Scaglione M. Safety and efficacy of pulmonary vein isolation using a surround flow catheter with contact force measurement capabilities: A multicenter registry. J Cardiovasc Electrophysiol. 2017 Jul;28(7):762-767. doi: 10.1111/jce.13227. Epub 2017 Jun 21. PMID 28422368